CLINICAL TRIAL: NCT06862232
Title: Efficacy and Outcomes of Winograd, Birdflap, and Noel's Surgical Techniques in Ingrown Toenail Treatment: A Prospective Randomized Controlled Study
Brief Title: P : Ingrown Toenail Patient I : Bird Flap Surgery C : Noel Winograd Method O : Recurrence, Complications, Functional Outcome, Pain,
Acronym: ITN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya City Hospital (Other)
Responsible Party: Principal Investigator, Bilgehan OCAK, Principal Investigator, Kutahya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KutahyaCH
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Ingrown Toenail
Keywords: ingrown toenail; birdflap surgery; winograd; recurrence; noel's surgery
MeSH Terms: conditions — Nails, Ingrown; Recurrence

STUDY DESIGN:
Intervention Model Description: The study is designed as a parallel-group, randomized controlled trial, consisting of three independent groups, each undergoing a different surgical technique for the treatment of medially ingrown toenails. Patients will be assigned to one of the three groups using a pre-generated randomized allocation list, ensuring an unbiased distribution. Each group will receive only the designated surgical intervention, with no crossover between groups.
  The surgical procedures will be performed according to the assigned technique, and postoperative outcomes-including recurrence rates, complications, pain levels, and functional recovery-will be assessed by an independent, blinded evaluator, ensuring objectivity and minimizing potential bias in outcome assessment.
Who Masked: Participant, Outcomes Assessor
Masking Description: To further minimize potential bias, the decision regarding the necessity of surgical intervention will be made by a surgeon independent of the study investigator. This ensures that the operating surgeon does not influence patient selection or determine which surgical technique is applied to each patient.
  All postoperative outcomes, including recurrence rates, complications, pain levels, and functional recovery, will be assessed by a separate independent, blinded evaluator, ensuring an objective assessment of surgical efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Winograd "Bird Flap" Technique (Experimental): Modified Winograd "Bird Flap" Technique
  In the first group (n=36), the modified Winograd "Bird Flap" technique will be performed. Local anesthesia will be administered using a 1% lidocaine solution, applied at the base of the first toe, and a temporary tourniquet will be placed using a sterile glove. The procedure involves creating an incision resembling the contour of a sparrow's body, extending over the lateral nail bed and reaching the proximal germinal matrix and underlying bone tissue. The granulated and infected tissue will be excised entirely to ensure complete removal of the affected area. The wound will then be sutured using 3/0 prolene sutures to achieve optimal wound closure. This technique aims to preserve the nail bed while effectively addressing the recurrence risk associated with conventional Winograd procedures.
  Interventions: Procedure: Modified Winograd "Bird Flap" Technique
- Modified Noel Technique (Active Comparator): Modified Noel Technique
  In the second group (n=36), the modified Noel technique will be utilized. Following local anesthesia with 1% lidocaine solution and the application of a temporary tourniquet, an approximately 4-6 mm semi-elliptical incision will be made adjacent to the lateral borders of the nail bed to access the granulated tissue. Unlike the Bird Flap technique, this method preserves both the nail bed and the proximal germinal matrix, ensuring that only the inflamed soft tissue and granulated tissue are excised. The remaining tissue will be sutured subungually using 3/0 prolene sutures to facilitate proper healing and maintain the structural integrity of the nail. This technique is designed to minimize invasiveness while effectively managing infected and inflamed tissue.
  Interventions: Procedure: Modified Noel Technique
- Classic Winograd Technique (Active Comparator): Classic Winograd Technique
  In the third group (n=36), the classic Winograd technique, a widely used traditional surgical approach, will be performed. After administering 1% lidocaine solution for local anesthesia and applying a temporary tourniquet, a linear incision will be made to separate the nail bed from the soft tissue. The lateral edge of the nail bed and the germinal matrix will then be excised in a linear fashion, ensuring complete removal of the affected nail portion. The wound will subsequently be sutured using 3/0 prolene sutures. This method has been a standard approach for ingrown toenail surgery and is associated with high recurrence prevention rates but also carries a risk of cosmetic and structural alterations in the nail.
  Interventions: Procedure: Classic Winograd Technique

INTERVENTIONS:
Procedure: Modified Winograd "Bird Flap" Technique — In the first group (n=36), the modified Winograd "Bird Flap" technique will be performed for medially ingrown toenails. Local anesthesia with 1% lidocaine will be administered at the base of the first toe, and a temporary tourniquet will be applied using a sterile glove to minimize bleeding.
  This technique modifies the Winograd method, optimizing functional and cosmetic outcomes while reducing recurrence rates. A sparrow-shaped incision will be made, encompassing the lateral nail bed, proximal germinal matrix, and underlying bone tissue, improving surgical access while preserving the healthy nail structure.
  Granulated and infected tissue will be excised completely down to the periosteum to prevent recurrence. The wound will be sutured using 3/0 prolene sutures, ensuring optimal healing and minimal scarring. This method aims to reduce pain, shorten recovery time, and improve patient satisfaction compared to traditional approaches.
  Arms: Modified Winograd "Bird Flap" Technique
Procedure: Classic Winograd Technique — The classic Winograd technique, a widely used traditional surgical approach, will be performed. Local anesthesia with 1% lidocaine will be administered, and a temporary tourniquet will be applied. A linear incision will be made to separate the nail bed from the soft tissue, followed by the excision of the lateral nail bed and germinal matrix in a linear fashion to ensure complete removal of the affected nail portion. The wound will then be sutured using 3/0 prolene sutures.
  This method is a standard approach for ingrown toenail surgery, offering high recurrence prevention rates but carrying a risk of cosmetic and structural nail alterations.
  Arms: Classic Winograd Technique
Procedure: Modified Noel Technique — Local anesthesia with 1% lidocaine will be administered, and a temporary tourniquet will be applied. A 4-6 mm semi-elliptical incision will be made adjacent to the lateral borders of the nail bed to access the granulated tissue.
  Unlike the Bird Flap technique, this method preserves both the nail bed and proximal germinal matrix, ensuring that only the inflamed soft tissue and granulated tissue are excised. The remaining tissue will be sutured subungually using 3/0 prolene sutures, promoting proper healing and maintaining the nail's structural integrity. This technique is designed to be less invasive while effectively treating infected and inflamed tissue.
  Arms: Modified Noel Technique

SUMMARY:
The treatment of ingrown toenails is highly diverse, with numerous surgical techniques described in the literature alongside conservative approaches. The primary goals of all these surgical methods are to reduce recurrence rates, improve patients' quality of life, and achieve favorable cosmetic outcomes. In this study, we aim to compare the recently introduced Bird Flap, a modified Winograd technique, with Noel's technique and the classic Winograd method in terms of recurrence rates, patient quality of life, cosmetic outcomes, and postoperative pain.

DETAILED DESCRIPTION:
Comparison of Surgical Techniques for Medially Ingrown Toenails: A Prospective Randomized Study

Introduction:

Medially ingrown toenail (Onychocryptosis) is a common foot condition that significantly affects patients by causing pain and discomfort, particularly while walking or wearing shoes. The condition is characterized by localized inflammation and bacterial infection around the nail bed, leading to purulent discharge. Patients with ingrown toenails are classified using the Hefetz classification system.

The treatment options for ingrown toenails are diverse, including both conservative and surgical approaches. The primary objectives of surgical interventions are to reduce recurrence rates, improve patient quality of life, and achieve optimal cosmetic outcomes. In this study, we aimed to compare the recently introduced Bird Flap (a modified Winograd technique), Noel's technique, and the classic Winograd method in terms of recurrence rates, patient-reported quality of life, cosmetic appearance, and postoperative pain.

Methods:

This study included three different surgical techniques applied to three separate patient groups.

* Group 1 (n=36): Patients underwent the modified Winograd "Bird Flap" technique, which involves an incision resembling the contour of a sparrow's body. Through this approach, the lateral nail bed, proximal germinal matrix, and granulation/infected tissue down to the bone were excised and subsequently sutured using prolene.
* Group 2 (n=36): Patients underwent the modified Noel technique, which involved a 4-6 mm semi-elliptical incision adjacent to the lateral margins of the nail bed, targeting the granulated tissue. Unlike the Bird Flap technique, this approach preserved the nail bed and proximal germinal matrix, with only the inflamed soft tissue and granulated tissue excised. The wound was then sutured subungually using prolene.
* Group 3 (n=36): Patients underwent the classic Winograd technique, which is the traditional method for ingrown toenail surgery. A linear incision was made to separate the nail bed from the soft tissue, followed by excision of the lateral edge of the nail bed and the germinal matrix in a linear fashion. The wound was then sutured accordingly.

Postoperative Follow-up and Outcome Measures:

All patients had their sutures removed on postoperative day 20 and were evaluated at 1-month, 2-month, and 3-month follow-ups.

* Primary Outcome: Recurrence rate
* Secondary Outcomes: Healing time, complications (bleeding, infection, wound site problems), and overall recovery and personal cosmetic satisfaction
* Pain, functional impact, and quality of life were assessed using the European Quality of Life Instrument (EuroQol) test.

This structured comparison provides insight into the effectiveness of these three distinct surgical approaches in managing medially ingrown toenails, with an emphasis on clinical and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of ingrown toenail (onychocryptosis)
* Indication for surgical treatment

Exclusion Criteria:

* Presence of malignancy in the body
* Existence of foot deformities
* Presence of pincer nail deformity
* History of drug allergy
* Presence of active infection in the body
* Diabetic neuropathy or necrotic foot ulcers
* Pregnancy
* History of prior foot or ankle surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Reccurence | six months
  The regrowth of the toenail towards the skin and/or soft tissue, leading to the recurrence of preoperative symptoms, characterized by pain, inflammation, and discomfort, occurring at any time within the first six months postoperatively.

SECONDARY OUTCOMES:
Recovery Time | 6 months
  Time to Resume Wearing Normal Footwear and Return to Work Duration
Complication | six months
  Severe pain, infection, bleeding, or wound care complications requiring hospital or physician intervention.
Life Qualty Assesment | six months
  Assessment of Pain, Functional Status, and Quality of Life using the EuroQol 5-Dimension 5-Level Scale (EQ-5D-5L). The EQ-5D-5L index score ranges from 0 to 1.000, with higher scores indicating better quality of life. Assessments will be conducted at 1-month, 2-month,3 months and 6-month follow-ups.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya City Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All participant will be share in epicollect5 and take all personal information and take a photo of toenail in both coronal and axial view
Supporting Information: Study Protocol, CSR
Time Frame: it will be available as long as study goes on
Access Criteria: all researchers https://five.epicollect.net/myprojects/my-thesis-about-ingrown-toenail
URL: https://five.epicollect.net/myprojects/my-thesis-about-ingrown-toenail

REFERENCES:
- [Background] Shang X, Jin Y, Meng X, Zhu H, Sun X, Xue Y, Rui Y. A novel modified Winograd surgical tricks and tips with a "bird flap" for the treatment of ingrown toenails. Foot Ankle Surg. 2023 Jun;29(4):361-366. doi: 10.1016/j.fas.2023.03.004. Epub 2023 Mar 15. PMID 36964004
- [Background] Dabrowski M, Litowinska A. Recurrence and satisfaction with sutured surgical treatment of an ingrown toenail. Ann Med Surg (Lond). 2020 Jun 26;56:152-160. doi: 10.1016/j.amsu.2020.06.029. eCollection 2020 Aug. PMID 32637092
- [Background] Livingston MH, Coriolano K, Jones SA. Nonrandomized assessment of ingrown toenails treated with excision of skinfold rather than toenail (NAILTEST): An observational study of the Vandenbos procedure. J Pediatr Surg. 2017 May;52(5):832-836. doi: 10.1016/j.jpedsurg.2017.01.029. Epub 2017 Jan 29. PMID 28190555